CLINICAL TRIAL: NCT00940706
Title: "Promotion of a Physically Active Lifestyle in Large Populations of Children and Teenagers With Cerebral Palsy in the Middle East"
Brief Title: Promotion of a Physically Active Lifestyle in Cerebral Palsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Fany Tusia, Proffesor Eli Lahat Primary Investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 481987103/09; MERC M29-023 (Other Grant/Funding Number: USA AID MERC M29-023)
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2009-07

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Activity monitoring; Treadmill; Group training; Physical active life style
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Test; Exercise; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical activity in groups (Experimental): Exercises of physical activity
  Interventions: Other: Physical activity in groups
- Activity monitoring with accelerometers (Experimental): Each subject will wear the accelerometer 24 hours a day for 4 days The activity will be recorded and analyzed
  Interventions: Behavioral: Monitoring physical activity
- Treadmill (Active Comparator): Treadmill with safety adaptations for handicapped persons
  Interventions: Device: TreadMill

INTERVENTIONS:
Device: TreadMill — Each subject will undergo 36 intervention sessions, 3 times a week, 12 weeks. Each session - up to 45 minutes
  TreadMill training: During each session the subject will first exercise with basic stretching and muscle strengthening and then walk on the treadmill. According to the subject's rate of improvement, a therapist will determine the rate of increase in the velocity and slope. The treating therapist will make a written report after each session.
  Other Names: TreadMill active focus physical training program
  Arms: Treadmill
Other: Physical activity in groups — Each subject will undergo 36 intervention sessions, 3 times a week, 12 weeks. Each session - up to 45 minutes.
  Activity Focus Training: this involves performing gross motor activities at exercise stations that involve repetitive, reciprocal and coordinated movements to facilitate strength and endurance conducted by physical therapists and instructing parents or other caregivers to be involved in the program. These activities are performed in a group, having a minimum of 6 children at one time.
  Other Names: Motor activity
  Arms: Physical activity in groups
Behavioral: Monitoring physical activity — Activity monitoring with accelerometers
  Other Names: Physical activity monitoring
  Arms: Activity monitoring with accelerometers

SUMMARY:
There is increasing evidence that physical activity during childhood and adolescence has an important impact on health and behavior outcomes. Lack of physical activity is currently a major concern for the total population and especially for children and adolescents. People with disabilities are at risk for the same health problems as the general population. Due to their disabilities, they have a higher risk for developing secondary conditions that may further affect their health and quality of life.The goals of this project are to develop and evaluate new approaches of treatment for children with cerebral palsy (CP) and to develop low cost tests for evaluating motor functions in natural environments.

The overall aim is to raise awareness of, and promote, a physically active lifestyle for Middle East teenagers with disabilities due to CP by means of a collaborative Jordanian-Israeli-Palestinian-Moroccan applied research project. Specific objectives include:

1. Evaluation of baseline levels of physical activity in large populations of children and teenagers with CP in the communities of the participating countries by long-term monitoring by accelerometers.
2. Conducting a randomized clinical trial to compare the efficacy of an "experimental" physical training program with a treadmill training program in two groups. The experimental training program is based on results of recent motor control studies, as well as the "motor learning" approach to facilitate transfer and retention of learned walking activities.
3. Disability Advocacy through dissemination of activity focus programs, raising awareness, making use of new technologies and enhancing and developing the skills and training of personnel working with populations with CP.
4. Continuing the expansion of collaborative research efforts pertaining to children and teenagers with physical disabilities between Arab countries and Israel through sharing of skills and knowledge by exchange visits, meetings and seminars and joint training, pediatric physiotherapists and physical educators.

DETAILED DESCRIPTION:
Stage I: Design A cross sectional research design.

Study participants for stage I: A total of 400 teenagers with CP will be monitored in this stage. All partners of this project will obtain approval for experiments on human subjects from their local committees. Each subject (or parents/guardians for the participation of minor subjects) will be able to sign an informed voluntary consent form, consistent with the Helsinki Declaration, after reading a detailed explanation and having an oral Q/A session with the investigator.

Recruitment: Prospective focused direct mailing or personal contacts will be initiated with the parents/guardians of children with CP who are ambulatory. Subsequent screening will be done by phone interview.

Participants at each center/country. 100 teenagers with CP, age 14-20 yr (50 age 14-17 yr and 50 age 18-20 yr). GMFCS levels II; III and IV.

Measurements:

Stage I:

The ActivePal accelerometer is a research instrument for long-term assessment of ambulatory activity during day-to-day life. Baseline functional status will be measured before interventions, including a completion of a socio-economical questionnaire.

Stage II: Randomized control trial of three training programs to improve the physical activity level and comparison between low and high costs interventions.

Study participants for Stage II. Thirty teenagers with CP at each center (total number of 120 at the four centers) will be matched according to age and GMFCS level (II and III) and randomly assign to one of three treatment programs. Subjects will be recruited from those in the first stage of the project. All partners of this project will obtain approval from their local committees. Each subject (or parents/guardians for the participation of a minor subject) will sign an informed voluntary consent form, consistent with the Helsinki Declaration, after reading a detailed explanation letter and having an oral Q/A session with the investigator.

Measurements:

2-Treadmill training measures will include total training time, step length, and with the split treadmill the velocity gap will also be recorded during each session 3-The gross motor function measure (GMFM) with dimensions D and E (standing, walking, running, jumping) will be used 4-Mechanical efficiency will be measured by the stair-climbing test.

Statistical analysis:

Repeated measures analysis of variance (ANOVA) will be used to determine the effects and compare the three treatment methods. The repeated measures factor will be the pre-post measurements and the grouping factors will be the functional levels (GMFCS) and treatment methods. Differences between pre-post measurements among the three methods will also be tested by one-way ANOVA. A p-value of < 0.05 will be considered significant.

ELIGIBILITY:
Stage II

Inclusion Criteria:

1. Diagnosis of cerebral palsy
2. Predominantly spastic type of CP with diplegia / tetraplegia
3. Age: 14 - 20 yr
4. GMFCS (gross motor function classification system) at levels II and III
5. A cognitive level sufficient to comprehend and cooperate in treatment and testing
6. No orthopedic surgery or other tone reduction intervention in last 6 months
7. Not a candidate for orthopedic surgical or other tone reduction intervention.

Exclusion Criteria:

1. Candidates for orthopedic surgical or other tone reduction procedures, e.g., botulin injections, baclofen pump interventions
2. Cannot cooperate in treatment or understand instructions
3. Uncontrolled convulsions if epileptic
4. Adolescents with progressive degenerative conditions of CNS or/and musculoskeletal system
5. Injury of lower extremity (reported fracture, sprain, strain) in the last 6 months
6. Orthopedic or neurological surgery in the last 12 months
7. Exercise induced asthma, cardiac problems and uncontrolled seizure disorders. Study Protocol. This stage will compare the efficacy of three training programs in increasing physical activity: a group physical activity program, a treadmill program and a split treadmill program.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The ActivPal is a research-grade instrument for long-term assessment of ambulatory activity during day-to-day life. The ActivPal is a highly accurate, unobtrusive instrument worn on the ankle. | stage I - 15 months stage II - 27 months

SECONDARY OUTCOMES:
The gross motor function measure (GMFM) with dimensions D and E (standing, walking, running, jumping) will be used. | before; after; 6 month after the comletion of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bar-Haim, PhD, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Bar-Haim S, Aviram R, Shkedy Rabani A, Amro A, Nammourah I, Al-Jarrah M, Raanan Y, Loeppky JA, Harries N. Effects of Exercise Interventions on Habitual Physical Activity and Sedentary Behavior in Adolescents With Cerebral Palsy. Pediatr Exerc Sci. 2019 Nov 1;31(4):416-424. doi: 10.1123/pes.2018-0254. Epub 2019 Jun 27. PMID 30922152
- [Derived] Shkedy Rabani A, Harries N, Namoora I, Al-Jarrah MD, Karniel A, Bar-Haim S. Duration and patterns of habitual physical activity in adolescents and young adults with cerebral palsy. Dev Med Child Neurol. 2014 Jul;56(7):673-80. doi: 10.1111/dmcn.12394. Epub 2014 Feb 10. PMID 24506509